CLINICAL TRIAL: NCT07239895
Title: Exploratory Study of Airway Basal Stem Cells on Treatment of Pediatric Bronchiolitis Obliterans
Brief Title: Treatment of Pediatric Bronchiolitis Obliterans by Airway Basal Stem Cells
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Regend Therapeutics (Industry)
Collaborators: Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO-V1.2
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Bronchiolitis Obliterans
Keywords: Airway Basal Stem Cells; Bronchiolitis obliterans; Bronchiolar Epithelium; Pedatric Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Airway Basal Stem Cells (Experimental)
  Interventions: Biological: Airway Basal Stem Cells

INTERVENTIONS:
Biological: Airway Basal Stem Cells — Airway Basal Stem Cells

SUMMARY:
Bronchiolitis obliterans (BO) is a chronic lung disease which was initiated with injury of the bronchiolar epithelium and resulted in nonuniform luminal obliteration or narrowing. Among children, the most common form of BO is post-infectious BO with a lack of treatment guidelines or standard therapy. In this study, an open, single-armed study is performed to preliminarily evaluate the safety and efficacy of airway basal stem cells on treatment of pediatric BO.

DETAILED DESCRIPTION:
The study is co-sponsored by Regend Therapeutics and Shanghai Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, aged between 28 days and 18 years;
* Diagnosed with bronchiolitis obliterans according to the guidelines;
* Meeting at least one of the following: FEV1 < 55% of predicted value; requiring continuous assisted mechanical ventilation or oxygen therapy;
* None of acute infections within the past four weeks;
* Tolerating bronchoscopy;
* The child and/or parent(s) provide informed consent, and are able to understand and adhere to scheduled visits, treatments, laboratory tests, and other study procedures.

Exclusion Criteria:

* Subjects with bronchiolitis obliterans syndrome (BOS) who are on a current cGVHD treatment regimen at screening.
* At the time of screening, subject who is positive in each of treponema pallidum antibody (TP-Ab), human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody test. Hepatitis B virus carriers with stable current condition can be enrolled. Cured hepatitis C patients with negative result in HCV ribonucleic acid (RNA) test can be enrolled as well.
* Subject who is assessed to have major lung diseases other than BO by investigators at screening or who has other severe systemic diseases within 6 months prior to screening and is considered to be unsuitable for this study by investigators.
* Presence of severe coagulation dysfunction at screening and may compromise the safety of bronchoscopy in the investigator's judgment.
* Subjects requiring long-term maintenance anticoagulant therapy or antiplatelet aggregation therapy, and for whom, in the investigator's assessment, the medication cannot be discontinued within a week prior to cell collection and infusion.
* Subjects with suicide risk or a history of psychiatric disorders at screening.
* Participation in another interventional clinical study within 3 months prior to screening.
* Poor compliance, making him or her difficult to complete the study.
* Subjects who is considered to be unsuitable for this study in in the opinion of the investigator.

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in clinical symptoms | 12 and 24 weeks after treatment
  Cough, wheezing, respiratory rate are included in clinical symptomes. Both status and frequency would be evaluated.
Changes in oxygen therapy | 24 weeks after treatment
  Oxygen saturation (SpO₂), oxygen therapy settings, and daily duration of oxygen therapy would be evaluated.

SECONDARY OUTCOMES:
Changes in general condition | 24 weeks after treatment
  Rate of weight gain, time of independent activity are evaluated as general condition.
Change in lung diffusing capacity for carbon monoxide (DLCO) from baseline | 12 and 24 weeks after treatment
  DLCO is a measure of the conductance of CO across the alveolar-capillary membrane and its binding with hemoglobin.
Change in forced expiratory volume in one second (FEV1) from baseline | 12 and 24 weeks after treatment
  FEV1 is the volume of breath exhaled with effort in one second.
Change in forced vital capacity (FVC) from baseline | 12 and 24 weeks after treatment
  FVC is the full amount of air that can be exhaled with effort in a complete breath
Change in high resolution computed tomography (HRCT) from baseline | 24 weeks after treatment
  HRCT scan is a type of CT scan that shows detailed pictures of lungs
Bronchiolitis Obliterans (BO) exacerbation | 24 weeks after treatment
  Frequency and severity of events will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No